CLINICAL TRIAL: NCT05655637
Title: Effects of Breathing Exercises Combined With Endurance and Strength Training on Dyspnea, Exercise Capacity and Quality of Life of Patients With Cystic Fibrosis.
Brief Title: Effects of Breathing Exercises Combined With Endurance and Strength Training in Patients With Cystic Fibrosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0342
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis Patients
Keywords: Cystic Fibrosis; Active cycle Breathing technique; 6 minute walk test; Borg scale; Quality of life
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): There will be one group, and study will be Quasi Experimental Study. Treatment will be given to all 28 participants, 3 sessions in a week for 4 weeks. Pre and Post treat-meant evaluation will be checked by CFQR+14. All patients will be treated with exercise program of Active cycle breathing techniques(ACBT), Pursed lip breathing, Endurance Exercise 20 to 30 min ( walking, cycling) and strength training with Thera-Bands (Bilateral arm raising, Bilateral knee extension). Exercise capacity will be measured with 6MWT. Dyspnea and fatigue will be measured with Borg scale.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — There will be one group, and study will be Quasi Experimental Study. Treatment will be given to all 28 participants, 3 sessions in a week for 4 weeks. Pre and Post treat-meant evaluation will be checked by CFQR+14. All patients will be treated with exercise program of Active cycle breathing techniques(ACBT), Pursed lip breathing, Endurance Exercise 20 to 30 min ( walking, cycling) and strength training with Thera-Bands (Bilateral arm raising, Bilateral knee extension). Exercise capacity will be measured with 6MWT. Dyspnea and fatigue will be measured with Borg scale.

SUMMARY:
Cystic fibrosis (CF) is a multi-system inherited disease. It's a common autosomal recessive illness. It mostly affects the lungs, liver, and pancreatic exocrine glands, as well as the intestines. The production of viscous mucus and an environment prone to chronic airway blockage. This allows harmful microorganisms to infect the lungs. The role of Exercise as a prognostic indicator or therapeutic aid is important in CF research around the world. The objective of this study is to find out the Effects of Breathing Exercises Combined with Endurance and Strength Training on Dyspnea and Quality of Life of patients with Cystic Fibrosis. It will be Quasi Experimental study. Treatment will be given to all participants 3 sessions in a week for 4 weeks. Pre and Post treat-meant evaluation will be checked by CFQ-R+14. All patients will be treated with exercise program of Active cycle breathing techniques(ACBT), Pursed lip breathing, Endurance Exercise 20 to 30 min ( walking, cycling) and strength training with Thera-Bands (Bilateral arm raising, Bilateral knee extension). Exercise capacity will be measured with 6MWT. Dyspnea and fatigue will be measured with Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-50 years
* Male and female both will be included
* clinically stable
* Shortness of breath on effort

Exclusion Criteria:

* smoking history >10 years
* clinical diagnosis of asthma
* Physical and psychological disability preventing participation
* medical condition which could place individuals at risk during exercise training

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
6-min walk test (6MWT) | 4 Weeks
  The 6-min walk test (6MWT) evaluates sub-maximal exercise responses. It's becoming more common in clinical studies, especially in situations of cardiopulmonary diseases like cystic fibrosis, where the patient's exercise ability and amount of physical activity are limited. It's used to assess functional capacity, conduct epidemiologic research, track the success of therapies, and predict morbidity and death for prognosis. The 6MWT is also regarded as a low-cost, easily repeatable outpatient test with high reliability and clinical use.
CFQ-R14+ | 4 Weeks
  Quality of life was measured by using the disease-specific health-related QoL questionnaire, CFQ-R 14+ The CFQ-R 14+ consists of 49 self-reported items within 12 domains: physical functioning , Vitality, emotional functioning, eating disturbances, treatment burden, general health perception, social functioning , body image, role limitations, weight problems, respiratory symptoms , digestive symptoms.
Borg Scale | 4 Weeks
  Borg scale is a validated indicator of the intensity of acute dyspnea. It ranges from 0 to 10 where a value of 0 represents "nothing at all", 5 is synonymous with "severe" and 10 signifies "maximal dyspnea".

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Bahria International Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mckoy NA, Wilson LM, Saldanha IJ, Odelola OA, Robinson KA. Active cycle of breathing technique for cystic fibrosis. Cochrane Database Syst Rev. 2016 Jul 5;7(7):CD007862. doi: 10.1002/14651858.CD007862.pub4. PMID 27378490
- [Background] Kapnadak SG, Dimango E, Hadjiliadis D, Hempstead SE, Tallarico E, Pilewski JM, Faro A, Albright J, Benden C, Blair S, Dellon EP, Gochenour D, Michelson P, Moshiree B, Neuringer I, Riedy C, Schindler T, Singer LG, Young D, Vignola L, Zukosky J, Simon RH. Cystic Fibrosis Foundation consensus guidelines for the care of individuals with advanced cystic fibrosis lung disease. J Cyst Fibros. 2020 May;19(3):344-354. doi: 10.1016/j.jcf.2020.02.015. Epub 2020 Feb 27. PMID 32115388
- [Background] Rand S, Prasad SA. Exercise as part of a cystic fibrosis therapeutic routine. Expert Rev Respir Med. 2012 Jun;6(3):341-51; quiz 352. doi: 10.1586/ers.12.19. PMID 22788948
- [Background] Pastre J, Prevotat A, Tardif C, Langlois C, Duhamel A, Wallaert B. Determinants of exercise capacity in cystic fibrosis patients with mild-to-moderate lung disease. BMC Pulm Med. 2014 Apr 30;14:74. doi: 10.1186/1471-2466-14-74. PMID 24884656
- [Background] Robinson KA, McKoy N, Saldanha I, Odelola OA. Active cycle of breathing technique for cystic fibrosis. Cochrane Database Syst Rev. 2010 Nov 10;(11):CD007862. doi: 10.1002/14651858.CD007862.pub2. PMID 21069699
- [Background] Ziegler B, Rovedder PM, Oliveira CL, de Abreu e Silva F, de Tarso Roth Dalcin P. Repeatability of the 6-minute walk test in adolescents and adults with cystic fibrosis. Respir Care. 2010 Aug;55(8):1020-5. PMID 20667149
- [Background] Quon BS, Wilkie SS, Ramsook AH, Schaeffer MR, Puyat JH, Wilcox PG, Guenette JA. Qualitative dimensions of exertional dyspnea in adults with cystic fibrosis. J Appl Physiol (1985). 2016 Aug 1;121(2):449-56. doi: 10.1152/japplphysiol.00391.2016. Epub 2016 Jun 16. PMID 27311438